CLINICAL TRIAL: NCT03225872
Title: Biology of Osteosarcoma (BOOST) Registry and Biobank
Acronym: BOOST
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2016NTLS073
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Bone cancer; Family-based study
MeSH Terms: conditions — Osteosarcoma; Bone Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The investigator will collect saliva and if available baby teeth. There will be no cost to you. If the investigator finds out that your sample doesn't have enough cells to be useful, the investigator may call you for an additional sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteosarcoma patients and family members: Osteosarcoma patients and family members

SUMMARY:
Osteosarcoma is very rare cancer of the bone. The investigator started the BOOST registry and biobank to make sure every patient has the opportunity to participate in research.

DETAILED DESCRIPTION:
Summary to include:

1. Samples of saliva, blood and/or other stored material such as slides or leftover diagnostic material. If available the investigator may ask you for deciduous (baby) teeth.
2. Questionnaire information, including health history, growth and development, physical activity and family medical history information.
3. If you have been diagnosed with a osteosarcoma or another condition the investigator is interested inthe investigator will ask you release medical record information relating to diagnosis and treatment of osteosarcoma, other cancers, blood disorders, and similar conditions. If this step applies to you then you will be asked to sign a separate form.
4. You may be asked to contact your biological parents and full biological siblings to ask them about participating in the study.
5. If you agree you may be contacted in the future. You will be able to decline any future information or studies at any point.

ELIGIBILITY:
Inclusion Criteria:

* Proband Inclusion criteria: A diagnosis or suspected diagnosis of osteosarcoma (ICCC 9180-9200)

Family member inclusion criteria: Biological parents and full biological siblings of a case diagnosed with osteosarcoma (ICCC 9180-9200)

Exclusion Criteria:

* Does not understand English.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Worldwide
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Determine if genes can determine osteosarcoma | Baseline
  To do this the investigator will compare the genes of people with osteosarcoma to the genes of people who do not have these conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Logan G. Spector, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided